CLINICAL TRIAL: NCT04897061
Title: Impact of Home Support on Quality of Post-operative Recovery After Major Pelvic Organ Prolapse Surgery
Brief Title: Caregiver Support and Post-operative Convalescence
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Ann Tran, MD, Assistant Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: IRB 20-01766
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Pelvic Organ Prolapse
Keywords: Prolapse; Same day discharge; Caregiver
MeSH Terms: conditions — Pelvic Organ Prolapse; Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants undergoing major pelvic organ prolapse surgery

SUMMARY:
This is a prospective cohort study designed to investigate the impact of home caregiver support on post-operative convalescence in patients undergoing same day discharge after major urogynecologic surgery. Questionnaires assessing post-operative convalescence will be distributed at several time points after surgery. The main hypothesis is that increased caregiver support in the post-operative period will improve post-operative convalescence of patients undergoing major urogynecologic surgery.

DETAILED DESCRIPTION:
Pelvic organ prolapse and incontinence surgery is now often done on an outpatient basis (also known as same day discharge surgery or SDD). While there are data to support the safety of this practice, little is known about the burden and demands of this practice on the patient and her support system/caregivers. Furthermore, there are no guidelines on requirements for assistance at home or what impact home caregiver support has on recovery. The study team is interested in investigating the spectrum of support that patients have at home in terms of caregivers such as family, friends, neighbors and how that may impact their recovery. The intervention for this study will be comprised of administering post-operative questionnaires that assess patients' post-operative convalescence and quantify the required or available caregiver support. The clinical outcome of interest is recovery as assessed by the validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* English speaking
* Successfully discharged on the day of surgery

Exclusion Criteria:

* Discharge to a nursing home, assisted living or rehabilitation facility.
* Dementia or altered mental status that would make recall of recovery process unreliable.
* Inability to access Internet or phone for study participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients are eligible to investigate post-operative recovery and convalescence after urogynecologic surgery.
Study Population: Women age 18 years or older undergoing major pelvic organ prolapse surgery (vaginal apical suspension, laparoscopic or robotic apical suspension, obliterative procedure) or minor prolapse or incontinence procedure with concomitant hysterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Recovery 15 (QOR-15) | Post-operative day 3, 7, 14, and 28
  Changes in Quality of Recovery 15 (QOR-15) scores based on a priori caregiver characteristics on post-operative days 3, 7, 14 and 28.
  QOR-15 is a 15 item instrument, full score range from 0 to 150, with higher score indicating better health outcomes.
Change in Post-discharge Surgical Recovery 13 (PSR-13) | Post-operative day 3, 7, 14, and 28
  Changes in Post-discharge Surgical Recovery 13 (PSR-13) scores based on a priori caregiver characteristics on post-operative days 3, 7, 14 and 28..
  The PSR scale is a 13 items instrument, full score range from 0-100, with higher score indicating better recovery.

SECONDARY OUTCOMES:
Change in Healthcare utilization composite score | Post-operative day 3, 7, 14, and 28
  Changes in a composite score comprised of healthcare utilization of phone calls, unanticipated office visits, and emergency department (ED) visits based on a priori caregiver characteristics on post-operative day 3, 7, 14, and 28.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Tran, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berg K, Idvall E, Nilsson U, Arestedt KF, Unosson M. Psychometric evaluation of the post-discharge surgical recovery scale. J Eval Clin Pract. 2010 Aug;16(4):794-801. doi: 10.1111/j.1365-2753.2009.01197.x. Epub 2010 Jun 14. PMID 20557414
- [Background] Kleinbeck SV. Self-reported at-home postoperative recovery. Res Nurs Health. 2000 Dec;23(6):461-72. doi: 10.1002/1098-240X(200012)23:63.0.CO;2-S. PMID 11130605
- [Background] Lassen PD, Moeller-Larsen H, DE Nully P. Same-day discharge after laparoscopic hysterectomy. Acta Obstet Gynecol Scand. 2012 Nov;91(11):1339-41. doi: 10.1111/j.1600-0412.2012.01535.x. Epub 2012 Oct 17. PMID 22924755
- [Background] Manohar A, Cheung K, Wu CL, Stierer TS. Burden incurred by patients and their caregivers after outpatient surgery: a prospective observational study. Clin Orthop Relat Res. 2014 May;472(5):1416-26. doi: 10.1007/s11999-013-3270-6. PMID 24005979
- [Background] Myles PS. Measuring quality of recovery in perioperative clinical trials. Curr Opin Anaesthesiol. 2018 Aug;31(4):396-401. doi: 10.1097/ACO.0000000000000612. PMID 29846193
- [Background] Wu CL, Berenholtz SM, Pronovost PJ, Fleisher LA. Systematic review and analysis of postdischarge symptoms after outpatient surgery. Anesthesiology. 2002 Apr;96(4):994-1003. doi: 10.1097/00000542-200204000-00030. No abstract available. PMID 11964610
- [Background] Berg K, Kjellgren K, Unosson M, Arestedt K. Postoperative recovery and its association with health-related quality of life among day surgery patients. BMC Nurs. 2012 Nov 13;11(1):24. doi: 10.1186/1472-6955-11-24. PMID 23148514
- [Background] Bouwsma EVA, Anema JR, Vonk Noordegraaf A, de Vet HCW, Huirne JAF. Using patient data to optimize an expert-based guideline on convalescence recommendations after gynecological surgery: a prospective cohort study. BMC Surg. 2017 Dec 6;17(1):129. doi: 10.1186/s12893-017-0317-8. PMID 29212492
- [Background] Carpenter JS, Heit M, Chen CX, Stewart R, Hamner J, Rand KL. Validating the Postdischarge Surgical Recovery Scale 13 as a Measure of Perceived Postoperative Recovery After Laparoscopic Sacrocolpopexy. Female Pelvic Med Reconstr Surg. 2017 Mar/Apr;23(2):86-89. doi: 10.1097/SPV.0000000000000352. PMID 28230616
- [Background] Chazapis M, Walker EM, Rooms MA, Kamming D, Moonesinghe SR. Measuring quality of recovery-15 after day case surgery. Br J Anaesth. 2016 Feb;116(2):241-8. doi: 10.1093/bja/aev413. PMID 26787793
- [Background] Dambi JM, Corten L, Chiwaridzo M, Jack H, Mlambo T, Jelsma J. A systematic review of the psychometric properties of the cross-cultural translations and adaptations of the Multidimensional Perceived Social Support Scale (MSPSS). Health Qual Life Outcomes. 2018 May 2;16(1):80. doi: 10.1186/s12955-018-0912-0. PMID 29716589
- [Background] Evenson M, Payne D, Nygaard I. Recovery at home after major gynecologic surgery: how do our patients fare? Obstet Gynecol. 2012 Apr;119(4):780-4. doi: 10.1097/AOG.0b013e31824bb15e. PMID 22433341
- [Background] Heit M, Carpenter JS, Chen CX, Stewart R, Hamner J, Rand KL. Predictors of Postdischarge Surgical Recovery Following Laparoscopic Sacrocolpopexy: A Prospective Cohort Study. Female Pelvic Med Reconstr Surg. 2020 May;26(5):320-326. doi: 10.1097/SPV.0000000000000599. PMID 29923843
- [Background] Kleif J, Waage J, Christensen KB, Gogenur I. Systematic review of the QoR-15 score, a patient- reported outcome measure measuring quality of recovery after surgery and anaesthesia. Br J Anaesth. 2018 Jan;120(1):28-36. doi: 10.1016/j.bja.2017.11.013. Epub 2017 Nov 22. PMID 29397134